CLINICAL TRIAL: NCT06743048
Title: Tissue Sparing Laser Assisted Penile Prosthesis Implantation
Brief Title: A Tissue Sparing, Laser Assisted Penile Prosthesis Implantation Technique
Acronym: TSLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adham ZAAZAA, Associate Professor Andrology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSLA_Implantation
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Erectile Dysfunction; Erectile Dysfunction Associated With Type 2 Diabetes Mellitus; Erectile Dysfunction Due to Arterial Disease; Erectile Dysfunction Due to Arterial Insufficiency; Erectile Dysfunction Due to Venous Disorder; Erectile Dysfunction Due to Neuropathy; Erectile Dysfunction Following Radical Prostatectomy
Keywords: Cavernosal tissue sparing laser assisted implantation
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TSLA Group (Other): Tissue Sparing Laser Assisted Penile Implantation
  Interventions: Procedure: Tissue Sparing Laser Implantation

INTERVENTIONS:
Procedure: Tissue Sparing Laser Implantation — A penile implant will be implanted using the cavernosal sparing technique and assisted by a laser fibre optic

SUMMARY:
A surgical technique using laser assisted penile prosthesis implantation

DETAILED DESCRIPTION:
A surgical technique using deep-red laser diode for visualization of the implantation track of the penile implant or Holium Laser for clearing the track whenever it is obstructed by fibrotic tissue.

ELIGIBILITY:
Inclusion Criteria:

* Men with ED not responding to medical treatment

Exclusion Criteria:

* Men with HBA1c more than 10

Ages: 21 Years to 81 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Males requiring penile implants
Enrollment: 7 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Successful Penile prosthesis implantation | 1 hour
  The penile implant is successfully implanted

CONTACTS AND LOCATIONS:
Locations (1):
- El Nada Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Sensitive data

REFERENCES:
- [Background] Zaazaa A, Mostafa T. Spontaneous Penile Tumescence by Sparing Cavernous Tissue in the Course of Malleable Penile Prosthesis Implantation. J Sex Med. 2019 Mar;16(3):474-478. doi: 10.1016/j.jsxm.2019.01.012. Epub 2019 Feb 14. PMID 30773500